CLINICAL TRIAL: NCT01595256
Title: Exploration the Effect of Individualized Home-based Walking Program on Muscle Strength and Fatigue in Patients With Colorectal Cancer Both During and After Treatment
Brief Title: Exploration the Effect of Walking Program in Patients With Colorectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 201109041RB
Record Dates: First submitted 2012-04-04; First posted 2012-05-10 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer,fatigue,6-minute walking test
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- walking group (Experimental)
  Interventions: Behavioral: muscular strength
- usual care (No Intervention)

INTERVENTIONS:
Behavioral: muscular strength — 12-week moderate intensity walking program
  Arms: walking group

SUMMARY:
The aims of this four-year study are to

1. explore the relationships between fatigue and muscle strength (i.e., upper limbs and lower legs)
2. comparison with the effects of 8-week, 12-week moderate intensity of walking program on muscle strength and fatigue.
3. develop a clinical guidelines of home-based walking program for patients with colorectal cancer receiving active treatment and survivors in Taiwan.
4. explore the relationships among the self-report fatigue intensity and metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Patients with colorectal cancer in receiving active treatment or completed treatment within 5years.
* Patients in Different Stages.
* Aged above 18.

Exclusion Criteria:

* KPS<60

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2011-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Exploration the Effect of Walking Program in Patients With Colorectal Cancer. | five-year study
  change of walking program on muscle strength and fatigue

CONTACTS AND LOCATIONS:
Overall Officials: Shiow-Ching Shun, PhD, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan